CLINICAL TRIAL: NCT01220609
Title: A Phase II Evaluation of Ixabepilone (NSC #710428) in the Treatment of Recurrent or Persistent Leiomyosarcoma of the Uterus
Brief Title: Ixabepilone in Treating Patients With Recurrent or Persistent Leiomyosarcoma of the Uterus Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02656; NCI-2011-02656 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000686644; GOG-0131H (Other: CTEP); U10CA027469 (NIH); U10CA180868 (NIH)
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Recurrent Uterine Corpus Sarcoma; Uterine Corpus Leiomyosarcoma
MeSH Terms: interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ixabepilone) (Experimental): Patients receive ixabepilone IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ixabepilone; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Ixabepilone — Given IV
  Other Names: BMS 247550; BMS-247550
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studying the side effects and how well ixabepilone works in treating patients with recurrent or persistent leiomyosarcoma of the uterus previously treated with chemotherapy. Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate (complete and partial responses by RECIST 1.1) of ixabepilone in patients with recurrent or persistent leiomyosarcoma of the uterus who have failed one previous chemotherapy regimen.

II. To determine the nature and degree of toxicity of ixabepilone as assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4 in this cohort of patients.

SECONDARY OBJECTIVES:

I. To determine the duration of progression-free survival (PFS) and overall survival (OS).

II. To determine the level of beta-III tubulin expression measured by IHC in women with leiomyosarcoma.

III. To determine if beta-III tubulin expression as measured by IHC predicts response to ixabepilone in women with leiomyosarcoma.

OUTLINE:

Patients receive ixabepilone intravenously (IV) over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed uterine leiomyosarcoma

  * Persistent or recurrent disease that is refractory to curative or established treatments
  * Histologic confirmation of the original primary tumor is required
* Measurable disease defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded)

  * Each lesion must be ≥ 10 mm by CT scan, MRI, or caliper measurement by clinical exam OR ≥ 20 mm by chest x-ray
  * Lymph nodes must be ≥ 15 mm in short axis by CT scan or MRI
* Must have ≥ 1 "target lesion" to assess response

  * Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence ≥ 90 days following completion of radiotherapy
* Not eligible for a higher priority GOG protocol, if one exists
* Must have had 1 prior cytotoxic regimen that included a taxane regimen for management of leiomyosarcoma

  * Single-agent or multi-agent therapy allowed
  * Patients who did not receive prior therapy with a taxane (e.g., docetaxel) must receive a second regimen that includes a taxane
* No known brain metastases
* GOG performance status 0-2
* Life expectancy > 6 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST ≤ 3 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Peripheral neuropathy (sensory or mother) ≤ grade 1
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception prior to and for the duration of study participation
* Free of active infection requiring antibiotics

  * Uncomplicated urinary tract infection allowed
* No other invasive malignancy except non-melanoma skin cancer or curatively treated localized cancer of the breast, head and neck, or skin that was completed more than 3 years ago and the patient remains free of recurrence or metastatic disease
* No history of a severe hypersensitivity reaction to agents containing Cremophor EL or its derivatives (e.g., polyoxyethylated castor oil)
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina
  * Cardiac arrhythmia
  * Psychiatric illness and/or social situations that would limit compliance with study requirements
* No concurrent amifostine or other protective agents
* Recovered from effects of recent surgery, radiotherapy, or chemotherapy
* At least 1 week since prior hormonal therapy

  * Hormonal therapy (cytotoxic or non-cytotoxic) not counted as prior regimen
* At least 3 weeks since any other prior therapy directed to the malignant tumor, including immunologic agents
* At least 4 weeks since prior radiation therapy
* One prior non-cytotoxic (biologic or cytostatic) regimen, administered as part of the previous cytotoxic regimen or in addition to it, allowed

  * Non-cytotoxic agents include, but are not limited to, the following:

    * Monoclonal antibodies
    * Cytokines
    * Small-molecule inhibitors of signal transduction
* More than 3 years since radiotherapy for localized cancer of the breast, head and neck, or skin provided patient remains free of recurrence or metastatic disease
* No prior ixabepilone
* No prior chemotherapy for any abdominal or pelvic tumor other than for the treatment of uterine leiomyosarcoma within the past 3 years
* Prior chemotherapy for localized breast cancer allowed provided it was completed more than 3 years ago and patient remains free of recurrent or metastatic disease
* No other concurrent investigational agents
* No concurrent strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, nefazodone, saquinavir, telithromycin, ritonavir, amprenavir, indinavir, nelfinavir, delavirdine, voriconazole, or grapefruit juice) or CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifampicin, rifabutin, phenobarbital, or St. John wort)
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-11; Primary Completion 2014-07 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Duska, Principal Investigator — NRG Oncology
Locations (72):
- United States (72):
  - Gynecologic Oncology Group of Arizona, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Cadence Cancer Center in Warrenville, Warrenville, Illinois
  - Saint Vincent Oncology Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Singing River Hospital, Pascagoula, Mississippi
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Ozark Health Ventures LLC-Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital - ProHealth Care, Waukesha, Wisconsin

REFERENCES:
- [Derived] Duska LR, Blessing JA, Rotmensch J, Mannel RS, Hanjani P, Rose PG, Dizon DS. A Phase II evaluation of ixabepilone (IND #59699, NSC #710428) in the treatment of recurrent or persistent leiomyosarcoma of the uterus: an NRG Oncology/Gynecologic Oncology Group Study. Gynecol Oncol. 2014 Oct;135(1):44-8. doi: 10.1016/j.ygyno.2014.07.101. Epub 2014 Aug 1. PMID 25091619

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixabepilone: Ixabepilone administered at 40 mg/m2 IV infusion over 3 hours on day 1 of a 21-day cycle until disease progression or adverse effects prohibit further treatment
Period: Overall Study
Arm/Group | Ixabepilone
Started | 26
Completed | 23 (Eligible and treated patients)
Not Completed | 3
Not completed — Ineligible-Wrong primary cancer site | 1
Not completed — Ineligible- Wrong cell type | 1
Not completed — Ineligible-Never treated | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Ixabepilone
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (7.1)
Age, Customized [Number; unit: participants]
  40-49 years | 5
  50-59 years | 12
  60-69 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Histologic Type [Number; unit: participants]
  Leiomyosarcoma | 22
  Carcinosarcoma, malignant mixed Mullerian tumor | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Complete and Partial Tumor Response by RECIST 1.1. RECIST 1.1 defines complete response as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and the disappearance of all non-target lesions and normalization of tumor marker level. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: Every other cycle for the first 6 months; then every 3 months thereafter; up to 5 years.
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone
Number analyzed (Participants) | 23
percentage of participants | 0 [0 to 100]

2. Primary Outcome: Frequency and Severity of Adverse Events as Assessed by NCI CTCAE v. 4.0
Time Frame: Every cycle until completion of study treatment up to 30 days after stopping study treatment
Population: Eligible and evaluable patients.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 4.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 4.0
- Grade 2 (CTCAE v 4.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 4.0
- Grade 3 (CTCAE v 4.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 4.0
- Grade 4 (CTCAE v 4.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 4.0
- Grade 5 (CTCAE v 4.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 4.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 4.0) | Grade 2 (CTCAE v 4.0) | Grade 3 (CTCAE v 4.0) | Grade 4 (CTCAE v 4.0) | Grade 5 (CTCAE v 4.0)
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23
Participants
  Leukopenia | 5 | 5 | 6 | 5 | 2 | 0
  Thrombocytopenia | 17 | 6 | 0 | 0 | 0 | 0
  Neutropenia | 8 | 4 | 4 | 3 | 4 | 0
  Anemia | 2 | 10 | 6 | 5 | 0 | 0
  Platelet count decreased | 17 | 6 | 0 | 0 | 0 | 0
  Nausea | 16 | 4 | 3 | 0 | 0 | 0
  Vomiting | 19 | 3 | 1 | 0 | 0 | 0
  Mucositis | 20 | 2 | 0 | 1 | 0 | 0
  Constipation | 15 | 7 | 1 | 0 | 0 | 0
  Diarrhea | 18 | 5 | 0 | 0 | 0 | 0
  Fatigue | 10 | 10 | 1 | 2 | 0 | 0
  Anorexia | 19 | 2 | 2 | 0 | 0 | 0
  Musculoskeletal/Connective tissue | 19 | 3 | 1 | 0 | 0 | 0
  Myalgia | 20 | 2 | 1 | 0 | 0 | 0
  Perpheral sensory neuropathy | 17 | 4 | 2 | 0 | 0 | 0
  Dizziness | 20 | 3 | 0 | 0 | 0 | 0
  Dyspnea | 19 | 2 | 1 | 1 | 0 | 0
  Alopecia | 13 | 4 | 6 | 0 | 0 | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression was based on RECIST 1.1. RECIST 1.1 defines progressive disease as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions or unequivocal progression of non-target lesions is also considered progression.
Time Frame: From study entry to disease progression, death or date of last contact, whichever occurs first, up to 5 years of follow-up.
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone
Number analyzed (Participants) | 23
months | 1.4 [1.2 to 1.6]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years of follow-up.
Population: Eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone
Number analyzed (Participants) | 23
months | 7.6 [4.5 to 13.6]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported.
Arm/Group | Ixabepilone
Serious Adverse Events (participants affected / at risk) | 9/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=23)
Dysphagia (Gastrointestinal disorders) | 1
Colonic Perforation (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Neutrophil Count Decreased (Investigations) | 3
Neoplasms Benign, Malignant And Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=23)
Anemia (Blood and lymphatic system disorders) | 21
Sinus Tachycardia (Cardiac disorders) | 1
Chest Pain - Cardiac (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
External Ear Inflammation (Ear and labyrinth disorders) | 1
Blurred Vision (Eye disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Bloating (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 3
Ileus (Gastrointestinal disorders) | 1
Oral Pain (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Edema Limbs (General disorders) | 3
Fatigue (General disorders) | 13
Fever (General disorders) | 1
Infusion Related Reaction (General disorders) | 1
Allergic Reaction (Immune system disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Weight Loss (Investigations) | 2
Weight Gain (Investigations) | 1
Platelet Count Decreased (Investigations) | 6
Neutrophil Count Decreased (Investigations) | 15
Blood Bilirubin Increased (Investigations) | 1
White Blood Cell Decreased (Investigations) | 18
Aspartate Aminotransferase Increased (Investigations) | 3
Alkaline Phosphatase Increased (Investigations) | 3
Alanine Aminotransferase Increased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal And Connective Tissue Disorder - (Musculoskeletal and connective tissue disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 7
Paresthesia (Nervous system disorders) | 3
Movements Involuntary (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 2
Urinary Frequency (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Bladder Spasm (Renal and urinary disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Scalp Pain (Skin and subcutaneous tissue disorders) | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 10
Thromboembolic Event (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less